CLINICAL TRIAL: NCT04041323
Title: Incidence and Outcomes of Acute Kidney Injury in Postoperative ICU Patients - a Retrospective Data Analysis
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, PD Peter Faybik, MD, Principal Investigator, Medical University of Vienna
Other Study IDs: EK Nr. 1419/2019
Record Dates: First submitted 2019-07-30; First posted 2019-08-01 (Actual); Last update posted 2021-11-30 (Actual); Status verified 2021-11

CONDITIONS: Acute Kidney Injury; ICU; Postoperative Patients
Keywords: AKI; KDIGO; ICU; postoperative
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Acute kidney injury (AKI) is a common complication in critically ill patients. Based on the sensitive KDIGO criteria, the incidence of AKI on ICU varies between 30-60 %. These large variations of incidence of AKI are due to different baseline characteristics of studied patients, the length of observation period, use of creatinine criteria only or use of creatinine and urine output criteria. Furthermore, back estimation of baseline creatinine instead of measured creatinine in patients with missing laboratory values may lead to overestimation of AKI severity and outcomes. Major surgery, trauma, infection, sepsis or a complication of severe illness can lead to an abrupt decrease in glomerular filtration in critically ill patients. Such episode of AKI is associated with short term adverse effects such as fluid overload, electrolyte imbalance, acid-base derangements, immune dysfunction, coagulation abnormalities and alterations in mental status. Additionally, AKI in critically ill patients leads to prolonged ICU length of stay, increase in morbidity and mortality as well as higher costs. Multiple large studies found, after correction for potential confounders, that AKI was independently associated with worse outcomes. Moderate and severe AKI stages were associated with 2.9 - 6.9 fold increased in-hospital mortality (3). Increasing AKI severity in ICU patients was not only associated with increased mortality, AKI patients had also worse renal function at the time of hospital discharge. The individual condition leading to AKI in combination with increased susceptibility to AKI may significantly influence outcome. Indeed, current data from many studies show that mortality from AKI differs in various clinical settings.

However, there are not enough data on different types of surgery and their effect on AKI yet. The aim of our epidemiological study is to investigate the occurrence and outcomes of AKI in different types of surgery in postoperative ICU patients at the Vienna General Hospital.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* postoperative ICU admission
* preoperative serum creatinine within 2 weeks prior surgery

Exclusion Criteria:

* age < 18 years
* no surgery prior to ICU admission
* renal transplantation prior ICU admission
* chronic renal replacement therapy
* peritoneal dialysis
* missing preoperative serum creatinine within 2 weeks prior surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: retrospective data analysis of postoperative ICU patients admitted to anaesthesiological and surgical ICUs of the General Hospital Vienna, Austria between January 1, 2016 and December 31, 2018.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Actual)
Dates: Start 2019-06-13 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
28 day mortality | 28 days
  primary outcome is the 28-day mortality in different stages of AKI according to KDIGO criteria in patients admitted in the ICU after surgery.

SECONDARY OUTCOMES:
ICU length of stay | 1 year
  secondary outcomes are length of stay in the ICU, receipt and duration of mechanical ventilation, receipt and duration of renal replacement therapy and 1- year all-cause mortality
receipt and duration of mechanical ventilation | 1 year
receipt and duration of renal replacement therapy | 1 year
1-year all cause mortality | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No